CLINICAL TRIAL: NCT01657708
Title: Implementation of Shared Decision Making Model in Psychiatric Rehabilitation Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SHA-0008-12
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Shared Decision Making With Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (1):
- Shared Desicion Making Model (Other)
  Interventions: Other: Shared Decision Making

INTERVENTIONS:
Other: Shared Decision Making

SUMMARY:
Background:

Shared Decision Making (SDM) refers to a process of health care delivery in which practitioners and clients seeking help with decisions, collaborate to access relevant information and enable client-centered selections of health care resources (1, 2). SDM leads to better treatment adherence and outcomes for people with a medical problem (3). SDM principles have previously been used in psychiatry to improve antipsychotic and antidepressant medication adherence (4, 5); however, these principles have yet to be applied to psychiatric rehabilitation (6).

The current research uniquely aims to test the development and implementation of a SDM intervention for people with psychotic spectrum disorders (e.g., schizophrenia and affective disorder) during the referral process to psychiatric rehabilitation services. The study will be conducted this year using a randomly selected sample from the population of people with psychotic spectrum disorders hospitalized in SHALVATA psychiatric hospital in Israel. It aims to facilitate better treatment and rehabilitation outcomes. It has received the support and approval of the Mental Health Division of the Ministry of Health (MOH) in Israel, the institutional review board (IRB) by the university of Haifa, Israel and a Helsinki committee approval by SHALVATA psychiatric hospital and the MOH in Israel.

References

1. Charles C, Gafni A, Whelan T. Shared decision-making in the medical encounter: What does it mean?(or it takes at least two to tango). Soc Sci Med. 1997;44(5):681-92.
2. Adams JR, Drake RE. Shared decision-making and evidence-based practice. Community Ment Health J. 2006;42(1):87-105.
3. Joosten EAG, DeFuentes-Merillas L, De Weert GH, Sensky T, Van Der Staak, C. P. F., De Jong, C. A. J. Systematic review of the effects of shared decision-making on patient satisfaction, treatment adherence and health status. Psychother Psychosom. 2008;77(4):219-26.
4. Hamann J, Cohen R, Leucht S, Busch R, Kissling W. Do patients with schizophrenia wish to be involved in decisions about their medical treatment? Am J Psychiatry. 2005;162(12):2382.
5. Hamann J, Langer B, Winkler V, Busch R, Cohen R, Leucht S, et al. Shared decision making for in-patients with schizophrenia. Acta Psychiatr Scand. 2006;114(4):265-73.
6. Drake RE, Deegan PE, Rapp C. The promise of shared decision making in mental health. Psychiatr Rehabil J. 2010;34(1):7-13.

ELIGIBILITY:
Inclusion Criteria:

* adults (over age 18), with severe mental illness signed an informed consent

Exclusion Criteria:

* do not understand Hebrew did not sign an inform consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Adherence to psychiatric rehabilitation services | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata psychiatric hospital, Hod HaSharon, Israel